CLINICAL TRIAL: NCT05615688
Title: Pain Intensity Following the Placement of Orthodontic Separators in Healthy Volunteers and How it Correlates to Different Levels of Physical Activity?
Brief Title: Pain and Activity Levels After Orthodontic Separators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lina Sharab (Other)
Responsible Party: Sponsor-Investigator, Lina Sharab, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 55656
Record Dates: First submitted 2022-08-19; First posted 2022-11-14 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Dental Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: Elastomeric separators will be placed on the mesial and distal of lower first permanent molars for a total of four separators per subject.
  Activity monitors will be provided and participants instructed to wear 24/7 unless showering or swimming to measure and collect level of physical activity
  Baseline data will be collected via questionnaires that include: Medical History, Demographics, and Perceived Stress Scale.
  Subjects will also complete a Recurrent Questionnaire at 2-4 hrs post placement and every evening for days 2-7 to report Pain Intensity using a Visual Analog Scale
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Orthodontic Separators Placed (Experimental): Elastomeric separators will be placed on the mesial and distal of the lower first permanent molars for a total of four separators per subject.
  Interventions: Procedure: Pain Intensity following Placement of Orthodontic Separators

INTERVENTIONS:
Procedure: Pain Intensity following Placement of Orthodontic Separators — Elastomeric separators will be placed on the mesial and distal of lower first permanent molars for a total of four separators per subject. Subjects will wear receive an activity monitor prior to placement of elastic separators and instructed to wear it 24/7 unless showering or swimming. Subjects will complete a recurrent Pain Scale Questionnaire 2-4 hrs after placement of elastics and every 24 hrs from day 2- 7.

SUMMARY:
The primary aim of this study is to evaluate the reported pain intensity following placement of Orthodontic separators on healthy volunteers aged 15-49 in relation to their recorded physical activity level.

Hypothesis 1: The investigators hypothesize that participants with higher daily step counts and physical activity levels will report significantly less pain intensity from orthodontic separators than their less active peers following separator placement. Null hypothesis is that participants with higher daily step counts will report the same pain intensity from orthodontic separators than their less active peers following separator placement

The secondary aim is to describe the course of pain, at 24 hr intervals, over the next seven days following separator placement.

Hypothesis 2: The investigators hypothesize that more physically active participants will report ratings of zero pain intensity faster (sooner) than their less active peers throughout the one week study. Secondary null hypothesis is that more physically active participants will report ratings of zero pain intensity at the same rate as their less active peers throughout the one week study.

DETAILED DESCRIPTION:
Acute pain or discomfort during orthodontic treatment is commonly reported. A study done in 2002 found that 87% of patients experienced pain after orthodontic visits. Additionally, "feeling pain" has been identified as the primary treatment concern for many patients prior to orthodontic treatment. More so, it can negatively affect patient compliance and attitude toward treatment.

Numerous studies have shown that pain varies in intensity and duration among orthodontic patients. The placement of orthodontic separators is a standard procedure to facilitate placement of orthodontic bands by creating a small amount of space between posterior teeth. Separator placement reliably produces acute discomfort to patients. Pain generated from orthodontic separator placement originates in the periodontal ligament (PDL) as compression forces are applied to the PDL unequally to open a small space (less than 0.5 mm) between the teeth. This compression triggers sterile necrosis or hyalinization in some areas of the PDL, leading to acute pain. The course of pain generated from orthodontic separators typically begins 4 hours after placement, reaching highest pain intensity approximately 24 hours after placement, and continuing to decrease in intensity until returning to pre-placement baseline after seven days.

Variation in reported pain intensity across orthodontic patients is of interest to any practitioner who desires to improve patient outcomes. In an attempt to enhance the orthodontist ability to understand pain and its predicting factors, researchers have examined pain from orthodontic treatment relative to patient demographics, personality traits, psychological factors, perceived need and attitude toward treatment, among others. Okeson asserts that pain is not directly related to the extent of tissue injury. Noxious stimuli originating in peripheral neurons (such is the case with separators) are subject to modulation at multiple levels through a complex central inhibitory system, where many other factors participate in decreasing or increasing the pain experience. Hence, an individual's emotional state, pain expectation and perception of control, as well as activities or distractions that will differ brain attention (Gate Control) can significantly influence the pain experience. Perceived stress, or the degree to which situations in an individual's life exceed their ability to cope, could be a good predictor of experienced pain. The Perceived Stress Scale is the most widely used screening form to evaluate perceived stress and asks subjects to recall the frequency of feeling overloaded and overwhelmed in the past month.

Recently, more attention has been given to the role of physical activity (PA) in reducing pain in patients that undergo orthodontic treatment. Physical activity has been shown to be an effective mediator of acute pain tolerance and pain sensitivity, an effect known as Exercise Induced Hypoalgesia (EIH). One study reported that a 1-mile run decreased pain intensity evoked from a weight being placed on the index finger. A similar decrease in pain response to pressure applied to the finger was found in subjects in another study who performed 30 minutes of aerobic exercise. It has also been demonstrated that exercise increased dental pain thresholds in response to electrical stimulation of the pulp. The exact mechanism involved in EIH remains elusive. Still, several pathways have been implicated including activation of the endogenous opioid pathway, increased Adrenocorticotropic Hormone release, and a conditioned pain the pain perceived in another area of the body.

Researchers have demonstrated that higher self-reported physical activity reduced the pain levels generated by placement of orthodontic separators when compared to patients with low physical activity. Self-reported measurements of physical activity carry limitations. The Physical Activity Questionnaire (PAQ) used in previous studies have demonstrated an only moderate correlation with direct activity observation (r=0.45), and with an activity monitoring device (r=0.57). The PAQ asks participants to report pain in the last seven days, and if given before treatment was performed, provides no data on physical activity during the week when subjects are experiencing pain. To further explore the correlation between physical activity and acute pain during orthodontic treatment, a more reliable measure of physical activity is warranted.

Actigraphy sensors provide an objective measure of physical activity. Actigraphy sensors include pedometers, which count steps over a defined time interval, and accelerometers, which measure acceleration in "activity counts" that are then extrapolated to the Metabolic Equivalent of Task (METS) to measure energy expenditure. No other paper has evaluated the effect of physical activity measured with pedometers on acute pain following separators placement during orthodontic treatment. Because not all patients experience pain at the same level, it would be beneficial for clinicians to identify which patients are likely to experience more intense pain before beginning treatment. To this end, the purpose of this study is to test the effect of physical activity measured by pedometer on acute pain produced by the placement of separators.

Protocol amended to include minors aged 15-17.

ELIGIBILITY:
Inclusion Criteria:

* Student, resident, or staff at the University of Kentucky
* Aged 15-49 at time of enrollment in the study
* Erupted permanent first and second molars with interproximal contacts
* Presence of antagonist teeth in the opposite arch with no open bite
* Voluntary participation in study
* Access to a smartphone, tablet, or computer
* Valid email address

Exclusion Criteria:

* Any chronic pain condition (examples include trigeminal neuralgia, migraines, fibromyalgia, arthritis, neuropathies)
* Current use of pain medication (analgesics, opioids, nerve pain medications) for any condition
* Clinically evident interproximal decay in the site where separators will be placed
* Missing teeth, variations in tooth anatomy, existing space, and or restorations that would keep separators from being placed or retained
* If you do not have access to a computer, smartphone, or tablet with internet access

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 94 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity | 7 days
  Subjects will be given an activity monitor to wear full time following the placement of the orthodontic spacers. They will report their level of pain to on a recurrent Pain Intensity questionnaire (using a Visual Analog Scale in REDCap) at 2-4 hrs after placement, and again at 24 hour intervals for the next 7 days following separator placement. The left of the digital Visual Analog Scale will be labeled "no pain" and the right will be labeled "worst pain imaginable". REDCap assigns a value of 0 on the left side of the scale and increased to100 on the right of the scale.

SECONDARY OUTCOMES:
Change in Proportion of patients reporting ZERO Pain over time | 7 days
  Subjects will be given an activity monitor to wear full time following the placement of the orthodontic spacers. They will report their level of pain on a recurrent Pain Intensity questionnaire (using a Visual Analog Scale in REDCap) at 2-4 hrs after placement, and again at 24 hour intervals for the next 7 days following separator placement. The left of the digital Visual Analog Scale will be labeled "no pain" and the right will be labeled "worst pain imaginable". REDCap assigns a value of 0 on the left side of the scale and increased to100 on the right of the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lina Sharab, DDS, MS, MSc, Principal Investigator — Assistant Professor, Orthodontics
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergius M, Berggren U, Kiliaridis S. Experience of pain during an orthodontic procedure. Eur J Oral Sci. 2002 Apr;110(2):92-8. doi: 10.1034/j.1600-0722.2002.11193.x. PMID 12013568
- [Background] Sergl HG, Klages U, Zentner A. Pain and discomfort during orthodontic treatment: causative factors and effects on compliance. Am J Orthod Dentofacial Orthop. 1998 Dec;114(6):684-91. doi: 10.1016/s0889-5406(98)70201-x. PMID 9844209
- [Background] Abu Alhaija ES, Aldaikki A, Al-Omairi MK, Al-Khateeb SN. The relationship between personality traits, pain perception and attitude toward orthodontic treatment. Angle Orthod. 2010 Nov;80(6):1141-9. doi: 10.2319/012710-59.1. PMID 20677967
- [Background] Beck VJ, Farella M, Chandler NP, Kieser JA, Thomson WM. Factors associated with pain induced by orthodontic separators. J Oral Rehabil. 2014 Apr;41(4):282-8. doi: 10.1111/joor.12144. Epub 2014 Feb 1. PMID 24483937
- [Background] Campos LA, Santos-Pinto A, Maroco J, Campos JADB. Pain perception in orthodontic patients: A model considering psychosocial and behavioural aspects. Orthod Craniofac Res. 2019 Aug;22(3):213-221. doi: 10.1111/ocr.12315. Epub 2019 May 15. PMID 31021044
- [Background] Rakhshan H, Rakhshan V. Pain and discomfort perceived during the initial stage of active fixed orthodontic treatment. Saudi Dent J. 2015 Apr;27(2):81-7. doi: 10.1016/j.sdentj.2014.11.002. Epub 2015 Jan 27. PMID 26082574
- [Background] Sandhu SS, Leckie G. Orthodontic pain trajectories in adolescents: Between-subject and within-subject variability in pain perception. Am J Orthod Dentofacial Orthop. 2016 Apr;149(4):491-500.e4. doi: 10.1016/j.ajodo.2015.10.020. PMID 27021453
- [Background] Sandhu SS, Sandhu J. Orthodontic pain: an interaction between age and sex in early and middle adolescence. Angle Orthod. 2013 Nov;83(6):966-72. doi: 10.2319/030113-174.1. Epub 2013 May 24. PMID 23705940
- [Background] Ngan P, Kess B, Wilson S. Perception of discomfort by patients undergoing orthodontic treatment. Am J Orthod Dentofacial Orthop. 1989 Jul;96(1):47-53. doi: 10.1016/0889-5406(89)90228-x. PMID 2750720
- [Background] Bondemark L, Fredriksson K, Ilros S. Separation effect and perception of pain and discomfort from two types of orthodontic separators. World J Orthod. 2004 Summer;5(2):172-6. PMID 15615136